CLINICAL TRIAL: NCT05735873
Title: The Clinical Impact of a Low-energy Diet on Medical Conditions Treated Within Bundled Payment Models: a Pilot Study
Brief Title: The Clinical Impact of Diet on Medical Conditions Treated Within Bundled Payment Models: a Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Leon Scott, Assistant Professor of Orthopaedic Surgery, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U13795
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee; Hypertension; Type 2 Diabetes; Obesity
Keywords: Caloric Restriction; Low energy diet; Value-based care
MeSH Terms: conditions — Osteoarthritis, Knee; Hypertension; Diabetes Mellitus, Type 2; Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Pilot study. Case series.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-energy diet arm (Experimental): Subjects who receive low-energy premade meals for three meals each day for 12 weeks.
  Interventions: Other: Low-energy diet

INTERVENTIONS:
Other: Low-energy diet — Twenty-one pre-made, low-energy meals delivered weekly to the subject for 12 weeks.

SUMMARY:
Diet interventions (e.g., low-energy diets) are recommended as a treatment for obesity, obese patients with osteoarthritis, hypertension (HTN), and type 2 diabetes (T2D). However, these diets are not a common part of the care plan partly because it is not financially feasible to discuss and offer them in medical offices reimbursed with the standard fee-for-service model. New reimbursement models, like value-based care (VBC), exist. It may be financially feasible to offer diet interventions, like premade and delivered meal plans to address these medical issues. This pilot study will help determine if a more extensive prospective study of the clinical effects of a delivered, premade low-energy diet (LED) on clinical markers of these disorders, as well as future cost-benefit analyses.

Methods: A case series of five obese subjects with knee osteoarthritis, HTN, and T2D receive a LED for 12 weeks. The primary outcome is the change in the Numeric Pain Rating Scale (NPRS) at 12 weeks. Secondary outcome measures include the change in other patient-reported outcomes between the start and end of the study, changes in weight, changes in measures of HTN and T2D, and the proportion of subjects using non-protocol interventions.

Hypothesis: Subjects randomized to the diet intervention will demonstrate a clinically significant improvement in NRPS score (2 points), a clinically significant weight reduction (15%), a 50% improvement in systolic and diastolic blood pressure, 1.0% reduction in Hemoglobin A1C levels (HgA1C), and lower utilization of non-protocol treatments at 12 weeks.

DETAILED DESCRIPTION:
Screening and Enrollment:

The subjects will be recruited from Vanderbilt University Medical Center's (VUMC) department of orthopaedics recent census of patients with the diagnosis codes for osteoarthritis (OA) of the knees (M17.11, M17.12, and M17.0), essential hypertension without heart failure (I11.9), type 1 diabetes (E10.) or type two diabetes controlled with insulin (E11.Z79.84). In addition, recruitment emails will be sent to VUMC employees using the VUMC email-based research notification system.

A Key Study Person (KSP) will conduct a screening call to review the inclusion and exclusion criteria. The potential subjects' charts will also be accessed to confirm age, sex, recent weight, and recent height. Eligible candidates would then meet a KSP for enrollment during a research visit.

Each patient will be asked to complete a questionnaire at the enrollment and 12-week research visits with the primary investigator. The questionnaire will be administered electronically into REDCap.

This questionnaire will survey the use of non-protocol interventions related to OA at any point during the intervention, such as (corticosteroid injection, viscosupplementation injection, platelet-rich plasma injection, weight loss prescription, or physical therapy) or in the week before completing the questionnaire (topical analgesic, oral analgesic, brace, or assistive walking device). The questionnaire will also include the following validated surveys for pain and function: Patient-reported Outcomes Measurement Information System Global Health Physical Function 10 (PROMIS-PF10), Numeric Pain Rating Scale (NRPS), Knee injury and Osteoarthritis Outcome Score (KOOS), and Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale.

In office measurements After enrollment, subjects will have their weight measured in their undergarments and an office gown. Their blood pressure will be collected with them seated on their left arm. Blood pressure will be measured using an automated sphygmomanometer (Philips Sure Signs VS4) three times with five minutes between measurements. The average systolic and diastolic measurements will be used as the research values.

A subject's height and weight will also be measured using an electronic scale (AWS SC2KGA ) while you are barefoot, wearing only a medical gown for full coverage. Your weight will be recorded as the weight of your body with the gown minus the weight of the gown alone.

These measurements will be collected at the enrollment and 12-week visits (research visits). Research visits will take place on Thursday afternoons at Vanderbilt Orthopaedics Franklin (VOF, 206 Bedford Way, Franklin, TN 37067)

Laboratories The Primary Investigator (PI) will collect blood for a HgbA1C at the research visits.

LED Meals Subjects will receive instructions on ordering their meals from the low-calorie meal service. Food will be available for pick up at VOF each Sunday between 4 pm and 6 pm for 12 weeks. Patients will receive reminders from a KSP to attend their research visits, complete their outcome questionnaires, and obtain other measurements and labs. Data from the questionnaire results will be de-identified. Then the PI will analyze the data, blind to the subjects and their interventions.

After enrollment, subjects can continue to seek care from their typical clinicians without instruction from the research team. There will not be any instruction from the research team to pursue, or avoid, care from their usual healthcare providers. The utilization of non-protocol interventions, like NSAID prescriptions or corticosteroid injections, will be monitored using the research visit questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 80 years of age
* Greater than, or equal to, four weeks of knee pain on the majority of days
* Weightbearing Xray within one year of enrollment demonstrating Kellgren Lawrence grade 1-4 changes
* Diagnosis of essential hypertension
* Diagnosis of type two diabetes.
* BMI >= 30kg/m2
* Consistent access to the internet
* Available on Thursdays for research visits
* Available each Sunday for 12 weeks between 4 pm and 6 pm to pick up the LED meals

Exclusion Criteria:

* Under 40 years of age
* Over 80 years of age
* Duration of symptoms less than four weeks
* Arthritis secondary to immune-mediated, infectious, or gout.
* Malignant hypertension
* Hypertension with heart-failure
* Secondary causes of hypertension
* Celiac disease, inflammatory bowel disease, gastroparesis, or other gastrointestinal disorders that can flare and reduce absorption.
* Tree nut or legume allergies
* Received any intraarticular knee injections in the past month.
* Using topiramate, phentermine, or glucagon-like peptide (GLP-1) agonists (e.g., semaglutide or dulaglutide)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to 12 weeks in Numeric Pain Rating Scale | Baseline to 12 weeks
  11-point scale that quantifies the amount of pain experienced over the preceding week. The score goes from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Change from Baseline to 12 weeks in Patient Reported Outcome Measurement Information System Physical Function10 | Baseline to 12 weeks
  A ten-question patient-reported outcome survey assesses how a subject's overall health impacts physical function. Each question has five responses, from 0 (no difficulty) to 5 (cannot do/unable to do). The sum of each response divided by the maximum score is reported as a percentage. 0% indicates the subject has no difficulty with global physical function; 100% indicates the subject is experiencing the maximum amount of limitation with physical function.
Change from Baseline to 12 weeks in Knee Osteoarthritis Outcome Score Subscales | Baseline to 12 weeks
  A 42-question Patient-reported outcome measures survey. It assesses the impact of knee osteoarthritis on five sub-scales: pain, symptoms, activities of daily living, recreation, and quality of life. A normalized score (100 indicating no pain and 0 indicating extreme pain) is calculated for each sub-scale.
Change from Baseline to 12 weeks in the Western Ontario and McMasters Osteoarthritis index | Baseline to 12 weeks
  A 24-question patient-reported outcome survey derived from the Knee Osteoarthritis Outcome Score reports a single score instead of sub-scales. Each question has five responses, from 0 (no difficulty) to 5 (extreme difficulty). The sum of each response divided by the maximum score is reported as a percentage. 0% indicates the subject is having no difficulty from osteoarthritis in the knee; 100% indicates the subject is experiencing the maximum amount of problem.
Change from Baseline to 12 weeks in Hemoglobin A1C | Baseline to 12 weeks
  A measure of the average blood glucose level over time
Change from Baseline to 12 weeks in systolic blood pressure | Baseline to 12 weeks
  A measure of the change in systolic blood pressure relative to a benchmark of 120 mm of Mercury
Change from Baseline to 12 weeks in diastolic blood pressure | Baseline to 12 weeks
  A measure of the change in diastolic blood pressure relative to a benchmark of 80 mm of Mercury

IPD SHARING:
Plan to Share IPD: No